CLINICAL TRIAL: NCT05754944
Title: Impact and Prevalence of PAD on Cancer Patients at High-risk for PAD Going to Surgery
Brief Title: Study of Peripheral Arterial Disease (PAD) in People With Cancer Who Will Be Having Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: BMS Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22-326
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease (PAD) in Cancer Patients
Keywords: Peripheral arterial disease (PAD); Cancer patients; 22-326
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients having surgery: This is a prospective cohort study where patients who are 65 years or older with either a history of diabetes (requiring medication or insulin) or smoking history (current smoker, smoker within the last 15 years, or ≥ 20 year pack history), facing major head and neck, thoracic, abdominal, or pelvic surgery will be screened for PAD with an ABI/TBI to establish prevalence and to compare prevalence among races to meet
  Interventions: Diagnostic Test: ABI/TBI; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: ABI/TBI — ABI/TBI to be performed after surgery while patient is still admitted at the hospital.
Other: Questionnaires — PAD symptoms questionnaire to be administered at baseline before surgery. mLEFS (included in PAD symptoms questionnaire) and WIQ to be administered at baseline before surgery. mLEFS and WIQ will be administered 1 month, 3 months, 6 months after surgery and every 6 months after that for a goal of at least 1 year.

SUMMARY:
Researchers are studying whether people with risk factors for blood circulation disease have a condition called peripheral arterial disease (PAD). People with PAD have poor blood circulation because of narrowing or blocks in blood vessels caused by fat or calcium deposits (atherosclerosis). The study researchers think that PAD may lead to worse outcomes in cancer treatment, but people with cancer are not routinely tested for the disease.

The purpose of this study is to find out how common PAD is among people with cancer who have risk factors for blood circulation disease, and to compare how often PAD is diagnosed in different racial groups

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who are ≥ 65 years old
* Either diabetes (on medication or insulin) or smoking history (current smoker, smoking within the last 15 years, ≥ 20 pack years)
* Patients who are scheduled for major head and neck, thoracic, abdominal, or pelvic surgery requiring at least a 2-day admission
* Ambulatory
* ≥ 6 month life expectancy as determined based on clinical judgement by the treating physician. If treating clinician does not confirm life-expectancy ≥ 6 months, will calculate Lee Schoenberg Index using ePrognosis.ucsf.edu.

Exclusion Criteria:

* Hospice patient, patient with a DNR order
* Non-ambulatory, wheelchair/bed bound
* < 6 month life expectancy based on the clinical judgement by the treating physician

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 65 years or older with either diabetes (requiring medication or insulin) or a smoking history (current smoker, smoker within the last 15 years, ≥ 20 year pack history), facing major head and neck, thoracic, abdominal, or pelvic surgery requiring at least at 2-day admission.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
prevalence of PAD in cancer patients at high-risk for PAD going to surgery | 1 year
  Completion of ABI/TBI to be able to assess prevalence of PAD

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Bryce, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm